CLINICAL TRIAL: NCT06411587
Title: Analysis of the Correlation Between Ultrasound Imaging and Functional Parameters in the Medial Gastrocnemius Muscle in Post-stroke Patients With Spasticity in the Lower Limb
Acronym: US-function
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Professor and PhD, Universidad de Zaragoza
Other Study IDs: US-function
Record Dates: First submitted 2024-03-08; First posted 2024-05-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Spasticity, Muscle
Keywords: Stroke; Ultrasound imaging; Spasticity, muscle; Function
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with stroke: Patients with a chronic stroke and spasticity in the ankle flexors muscles.
  Interventions: Diagnostic Test: Ultrasound imaging and functional assessment
- Patients without stroke: Patients without stroke were matched with those with stroke based on age and sex.
  Interventions: Diagnostic Test: Ultrasound imaging and functional assessment

INTERVENTIONS:
Diagnostic Test: Ultrasound imaging and functional assessment — Participants in this study will undergo two types of assessments: capturing muscle images using ultrasound and evaluating their function through clinical scales.

SUMMARY:
The goal of this observational study is to understand the impact of spasticity on muscle changes and functional performance in stroke patients with lower limb spasticity in comparison to non-stroke individuals. The main questions it aims to answer are:

* How does spasticity affect muscle changes and lower limb functional performance in stroke patients?
* How do structural and textural parameters in ultrasound images differ between spastic stroke patients and non-stroke individuals?

Participants will undergo ultrasound evaluation of their leg muscles to measure structural and textural parameters. They will also take part in functional assessments to assess their performance in activities related to lower limb mobility.

Researchers will compare the structural and textural ultrasound parameters between stroke patients and non-stroke individuals to determine any notable differences. The study aims to identify the relationship between muscle changes, spasticity, and functional performance in stroke patients.

DETAILED DESCRIPTION:
Cerebrovascular Accident (CVA) or stroke is one of the leading causes of morbidity and disability worldwide. Spasticity is a common complication in patients with CVA, affecting between 43.2% and 49.5% of patients in the first six months. It can interfere with movement and cause discomfort, pain, joint contracture, and abnormal limb posture. Ankle spasticity is particularly problematic for gait recovery.

Computed tomography (CT) and magnetic resonance imaging (MRI) are considered the gold standard for measuring muscle mass, but their use is not practical due to patient discomfort, radiation exposure, and high costs. Ultrasound is presented as an effective and low-cost tool for evaluating muscle tissues.

Previous research has analyzed architectural changes in spastic muscles in hemiplegic patients and found conflicting results regarding muscle thickness and fascicle length. Further studies are needed to better understand the relationship between muscle changes and weakness, spasticity, and functional performance of the lower limbs.

This study aims to analyze the relationship between muscular architecture and echotexture parameters, and the functional parameters of the medial gastrocnemius muscle in patients with spasticity in the lower limb after a stroke and compare them with non-stroke subjects.

Comparing the affected side with the supposedly healthy side of stroke patients will allow for a better understanding of the structural changes that occur on both sides.

Studying structural changes in patients with chronic spasticity after a stroke can help healthcare professionals better understand the impact of this condition on muscle function and develop personalized treatment plans. Ultrasound can be a useful tool to improve the effectiveness of rehabilitation interventions in stroke survivors.

ELIGIBILITY:
Group of patients diagnosed with ischemic or hemorrhagic stroke.

Inclusion Criteria:

* Age over 18 years
* Present spasticity in the plantar flexor muscles of the ankle as a result of a first unilateral ischemic or hemorrhagic stroke (excluding subarachnoid hemorrhage, as it is not truly a stroke) diagnosed by computed tomography or magnetic resonance imaging.
* Have more than 6 months of evolution since the onset of the cerebrovascular accident (chronic stroke).
* Degree of spasticity on the Modified Ashworth Scale (MAS): 1, 1+, 2, or 3.
* Be able to walk independently with or without assistance.

Exclusion Criteria:

* Other musculoskeletal or neurological disorders affecting the lower limb (bilateral stroke, peripheral neuropathy, peripheral nerve injury, myopathy, severe osteoarthritis, recent muscle injury, recent bone fracture, joint replacement, fixed contractures involving the affected leg, bone deformities of the lower limbs).
* Other neurological pathologies (e.g., ataxia or dystonia).
* Surgical intervention in the lower limb.
* Cognitive impairments that hinder study measurements.
* Other medical conditions that may interfere with data interpretation.

Group of non-stroke patients

Inclusion Criteria:

* Age over 18 years
* Be able to walk independently with or without assistance

Exclusion Criteria:

* Previous diagnosis of stroke.
* Presence of spasticity in any part of the body.
* Other musculoskeletal or neurological disorders affecting the lower limb (bilateral stroke, peripheral neuropathy, peripheral nerve injury, myopathy, severe osteoarthritis, recent muscle injury, recent bone fracture, joint replacement, fixed contractures involving the affected leg, bone deformities of the lower limbs).
* Other neurological pathologies (e.g., ataxia or dystonia).
* Surgical intervention in the lower limb.
* Cognitive impairments that hinder study measurements.
* Other medical conditions that may interfere with data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke group: patients diagnosed with ischemic or hemorrhagic stroke who follow the selection criteria.
  Non-stroke group: patients without a diagnosis of stroke matching with each member of the stroke group.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | Through study completion, an average of 1 year
  It is the distance between the superficial and deep layer of the fascia of the medial gastrocnemius. It is considered one of the 3 muscular architecture parameters that will be measured using ultrasound images collected with the Butterfly iQ+ portable device by Butterfly Network, Inc., a company located in the United Kingdom. The device is connected to a tablet from which the images are visualized and captured. For more information about the device, you can visit the following link: www.butterflynetwork.com/int/es-es/individual

SECONDARY OUTCOMES:
Fascicle length | Through study completion, an average of 1 year
  It is the estimation of the length of the muscle fiber, which is obtained by tracing a line that covers the length of the muscle fascicle between the deep and superficial aponeuroses.
Pennation angle | Through study completion, an average of 1 year
  It is the angle between the deep fascia and the line of the fascicle length.
Concurrence matrices | Through study completion, an average of 1 year
  Measures that describe the spatial distribution of gray levels in the texture of an ultrasound image. These matrices, also known as co-occurrence matrices, are used to analyze textural features and patterns in ultrasound images.
Degree of spasticity | Through study completion, an average of 1 year
  It will be measured using the Modified Ashworth Scale (MAS). The scale ranges from a minimum value of 0 to a maximum of 4, with 0 indicating no spasticity and 4 representing the most severe spasticity, characterized by complete rigidity.
Functional capacity | Through study completion, an average of 1 year
  Measured by Time Up and Go (TUG)
Functional capacity | Through study completion, an average of 1 year
  Measured by 10 Meter Walk Test (10MWT)
Muscle strength | Through study completion, an average of 1 year
  Maximum isometric contractions will be measured using dynamometry.
Contraction velocity, relaxation velocity, and shrinkage potential | Through study completion, an average of 1 year
  The Movement mode will be used to calculate these parameters simultaneously taken the force using dynamometry. This will allow correlating the Modo M with force.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero Gallego, Physical Therapist, Study Director — Universidad de Zaragoza
Locations (1):
- Universidad de Zaragoza, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The team is still figure it out what is the best way to share the information.